CLINICAL TRIAL: NCT03543709
Title: Evaluation of Fibromyalgia With Disease Activity and Clinical Findings in Women With Behçet's Disease in Province Bursa
Brief Title: Evaluation of Fibromyalgia With Disease Activity and Clinical Findings in Women With Behçet's Disease
Status: Completed | Type: Observational
Sponsor: Bursa Yuksek Ihtisas Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Koray Ayar, Assistant Professor, Bursa Yuksek Ihtisas Training and Research Hospital
Other Study IDs: 2011-KAEK-26/105
Record Dates: First submitted 2018-05-21; First posted 2018-06-01 (Actual); Last update posted 2019-02-06 (Actual); Status verified 2019-02

CONDITIONS: Behcet's Disease; Fibromyalgia
Keywords: Behcet's disease; Fibromyalgia; Disease activity
MeSH Terms: conditions — Behcet Syndrome; Fibromyalgia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Behcet and fibromyalgia: Women with Behcet's disease with fibromyalgia
  Interventions: Diagnostic Test: fibromyalgia 2013 criteria; Other: Behcet's disease current activity form
- Behcet: Women with Behcet's disease without fibromyalgia
  Interventions: Diagnostic Test: fibromyalgia 2013 criteria; Other: Behcet's disease current activity form

INTERVENTIONS:
Diagnostic Test: fibromyalgia 2013 criteria — Frequency of fibromyalgia will be investigated in women diagnosed with Behcet disease
Other: Behcet's disease current activity form — Disease activity will be investigated in women with Behçet's disease without fibromyalgia.

SUMMARY:
In the literature, the relationship between fibromyalgia and disease activity has been assessed in a few studies without discrimination between women and men.In this study, it was aimed to evaluate the relationship between fibromyalgia and disease activity in women with Behçet's disease.

DETAILED DESCRIPTION:
There are only a few studies in the literature evaluating the association of fibromyalgia with disease activity and clinical findings in Behçet's disease. In the literature, the relationship between fibromyalgia and disease activity has been assessed without discrimination between women and men. Behçet's disease is more active in men and fibromyalgia is more frequent in women. Evaluating the relationship between fibromyalgia and disease activity in Behçet's disease without gender discrimination may not be objective.There is not any study in literature evaluating relationship between fibromyalgia and disease activity in women with Behçet's disease.In this study, it was aimed to evaluate the relationship between fibromyalgia and disease activity in women with Behçet's disease.

ELIGIBILITY:
Inclusion Criteria:

* Women diagnosed with Behcet disease according to international study group criteria
* Patients older than 18
* Patients younger than 75

Exclusion Criteria:

* Participants which were previously diagnosed with diabetes mellitus
* Participants which were previously diagnosed with chronic renal failure
* Pregnant women

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women diagnosed with Behcet disease according to international study group criteria, between age 18-75, which are not pregnant and which were not previously diagnosed with diabetes mellitus or chronic renal failure.
Sampling Method: Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2018-06-11 (Actual); Primary Completion 2019-02-05 (Actual); Study Completion 2019-02-05 (Actual)

PRIMARY OUTCOMES:
Fibromyalgia 2013 criteria | 5 months
  Fibromyalgia 2013 criteria were derived from the 10-item symptom score from the Symptom Impact Questionnaire (SIQR) symptoms and the 28-area pain location inventory (PLI). If the patients PLI score is above 17 (range 0-28) and an SIQR symptom score is above 21 (range 0-50), the participant will be diagnosed with fibromyalgia

SECONDARY OUTCOMES:
Behcet's disease current activity form | 5 months
  Twelve items on the Behcet's disease current activity form, a potential unidimensional scale, will be used for the analysis as well as the two questions which assess disease activity from the patient's and clinician's perspective. These items are: a Likert scale, represented by 'smiley' faces ranging from very bad to very good, to indicate how the patient or the clinician felt the disease had been over the past 4 weeks, and the presence or absence (over the last 4 weeks prior to the clinic visit) of arthralgia, arthritis, diarrhoea, erythema nodosum, eye inflammation, genital ulcers, headaches, mouth ulcers, nausea/vomiting, new central nervous system involvement, new major vessel inflammation, and pustules.

CONTACTS AND LOCATIONS:
Locations (1):
- Koray, Bursa, Turkey (Türkiye)